CLINICAL TRIAL: NCT00083148
Title: Phase I Study of Irinotecan Followed by Capecitabine in Patients With Advanced Breast Carcinoma
Brief Title: Irinotecan and Capecitabine in Treating Women With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Tracey O'Connor, MD, Roswell Park Cancer Institute
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CDR0000363790; RPCI-RP-0221
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Irinotecan may help capecitabine kill more tumor cells by making tumor cells more sensitive to the drug.

PURPOSE: This phase I trial is studying the side effects and best dose of irinotecan and capecitabine in treating women with advanced breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of capecitabine and irinotecan in women with advanced breast cancer.
* Determine the degree of accumulation of cells in S-phase in tumor biopsies from patients treated with this regimen.
* Determine the dose-limiting toxicity and other major or unusual toxic effects of this regimen in these patients.
* Determine any antitumor activity of this regimen in these patients.
* Determine the pharmacokinetics of this regimen, including the active metabolite SN-38, in these patients.
* Correlate pharmacokinetic parameters of this regimen with the biological changes observed in these patients.
* Determine, preliminarily, the relationship of tumor response with modulation of S-phase in patients treated with this regimen.

OUTLINE: This is a dose-escalation study.

Patients receive irinotecan IV over 1.5 hours on days 1, 8, 22, and 29 and oral capecitabine twice daily on days 1-14 and 23-36. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of irinotecan and capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 8-37 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer not eligible for potentially curative therapy or studies of higher priority

  * Advanced disease
  * Tumor accessible to biopsy AND not irradiated
* Failed at least 1 prior chemotherapy regimen (not including adjuvant chemotherapy)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* AST ≤ 2 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN

Renal

* Creatinine ≤ 1.5 times ULN OR
* Creatinine clearance ≥ 50 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active uncontrolled bacterial, viral, or fungal infection
* No poor medical risk from non-malignant systemic disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* Prior irinotecan allowed
* Prior carboplatin allowed
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy except for small port radiotherapy for local control

Surgery

* More than 4 weeks since prior major surgery

Other

* No concurrent high-dose IV cyclosporine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2002-11; Primary Completion 2005-03 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey O'Connor, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Result] O'connor T, Rustum Y, Levine E, Creaven P. A phase I study of capecitabine and a modulatory dose of irinotecan in metastatic breast cancer. Cancer Chemother Pharmacol. 2008 Jan;61(1):125-31. doi: 10.1007/s00280-007-0456-1. Epub 2007 Apr 11. PMID 17426973